CLINICAL TRIAL: NCT02092792
Title: A PHASE I, OPEN-LABEL STUDY EVALUATING THE SAFETY AND TOLERABILITY OF ESCALATING DOSES OF DLYE5953A IN PATIENTS WITH REFRACTORY SOLID TUMORS
Brief Title: A Study Evaluating the Safety of Escalating Doses of DLYE5953A in Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29146
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Dose-Escalation Phase (Experimental)
  Interventions: Drug: DLYE5953A
- Dose-expansion cohort (Experimental)
  Interventions: Drug: DLYE5953A

INTERVENTIONS:
Drug: DLYE5953A — Escalating doses of DLYE5953A
  Arms: Dose-Escalation Phase
Drug: DLYE5953A — Administration of DLYE5953A at the recommended phase II dose (RP2D)
  Arms: Dose-expansion cohort

SUMMARY:
This is an open-label, multicenter, Phase I study to evaluate the safety, tolerability, and PK of escalating doses of DLYE5953A administered to patients with incurable, locally advanced, or metastatic solid malignancy that has progressed on standard therapy. The Phase I study consists of two stages: Stage 1 dose-escalation and Stage 2 expansion in selected patients. In Stage 1, a 3 + 3 dose-escalation design will be used to examine the safety, tolerability, and PK of increasing doses of DLYE5953A. In Stage 2, patients will be enrolled to further characterize the safety, tolerability, and PK of the proposed dose and schedule for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* ECOG performance status of 0 or 1
* Histologically or cytologically documented advanced or metastatic solid tumors for which established therapy either does not exist or has proven ineffective or intolerable
* Measurable disease by RECIST v1.1 with at least one measurable target lesion

Exclusion Criteria:

* Treatment with chemotherapy, hormonal therapy (except hormone replacement therapy, oral contraceptives), immunotherapy, biologic therapy, radiation therapy (except palliative radiation to bony metastases), or herbal therapy as cancer therapy within 4 weeks prior to initiation of DLYE5953A
* Oral kinase inhibitors approved by local regulatory authorities may be used within 2 weeks prior to initiation of DLYE5953A, provided that any clinically relevant drug-related toxicity has completely resolved and prior approval is obtained from the Medical Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | Days 1 to 21
Incidence of adverse events | Up to 32 months

SECONDARY OUTCOMES:
Total exposure of the drug, defined as the area under the concentration-time curve (AUC) | Up to 32 months
Incidence of anti-DLYE5953A antibodies | Up to 32 months
Objective response according to Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1 | Up to 32 months
Duration of objective response | Up to 32 months
Progression-free survival | Up to 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York